CLINICAL TRIAL: NCT06054737
Title: Effectiveness of the Spa Therapy Program of Royat in Chronic Venous Insufficiency
Brief Title: Chronic Venous Insufficiency and Balneotherapy
Status: Completed | Type: Observational
Sponsor: CEN Biotech (Industry)
Collaborators: TOWN HALL OF ROYAT (Unknown)
Responsible Party: Sponsor
Other Study IDs: C1688
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Venous Insufficiency (Chronic)(Peripheral)
Keywords: Spa therapy,; Balneotherapy; Chronic venous insufficiency; CVI; CVD
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SPA THERAPY PROGRAM: 3-week spa therapy program with Mineral Water of Royat in addition to standard of care for chronic venous insufficiency
  Interventions: Procedure: SPA THERAPY

INTERVENTIONS:
Procedure: SPA THERAPY — Balneotherapy program Four balneotherapy sessions per day, 6 days a week during 3 weeks
  The balneotherapy sessions included:
  * 10- minute walking session in a specially designed pool with tracks in semideep (80 cm) cool (30°C) water (training of muscle pump function under water compression);
  * 20-minute whirlpool bath session with automatic air or submarine bath if hypodermis (aimed at relaxation and mobilization of the superficial skin volume flow); followed by a 10-minute hydrojet bath (2 sessions) with customized underwater strong massaging jets (mobilization and softening of the sclerotic subcutaneous tissues);
  * Fresh thermal water compresses at 24°C. The cool temperature of the compresses also has an analgesic and decongestant effect. This treatment is carried out last and is followed by a rest for a total duration of 60 minutes
  Other Names: BALNEOTHERAPY THERAPEUTIC ORIENTATION PHLEBOLOGY

SUMMARY:
The aim of this clinical trial is to assess the efficacy of the balneotherapy program (therapeutic orientation: Phlebology) in terms of chronic venous disease improvement and related quality of life, in patients presented with advanced chronic venous insufficiency (i.e., with C4-C5 of severity classification).

The multicenter randomized controlled trial (RCT) "Thermes & Veines" that aimed at evaluating balneotherapy in patients with advanced chronic venous insufficiency is considered as the reference study. The French National Academy of Medicine encourages the re-use of data of published RCT when available. In this context, the current study is designed as a single-arm prospective study with indirect comparison using propension score. The Control group consists of the 197 patients which were allocated to the Control group of the "Thermes & Veines".

All patients enrolled in the current study benefit of 18-days of spa treatment with Mineral Water of Royat, and examination with vascular practitioner at enrollment and 6 months after the beginning of spa treatment.

DETAILED DESCRIPTION:
Chronic Vascular Disease (CVD) related quality of life and symptoms, as well as skin trophic changes from baseline are assessed at 6 months. Variations from baseline are compared in Control and Spa treatment groups. The indirect comparison methodology is based on the reuse of individual data from a "control" group and adjustment after calculating the propensity score.

ELIGIBILITY:
Inclusion Criteria:

* Primary or post-thrombotic CVD with confirmed diagnosis by by duplex ultrasound examination (last available exam);
* With CVI classified as C4a, C4b, or C5)
* Available for balneotherapy program within the 2 next months
* With health insurance affiliation.

Exclusion Criteria:

* Active venous thrombosis, recent or ongoing erysipelas, peripheral arterial pathology (ankle brachial index < 0.70).
* Walking difficulty
* Neurologic diseases of the lower limbs
* Presenting or likely to present a contraindication to thermal treatments, with planned surgery;
* Having already benefited from a thermal treatment whatever the indication during the last 6 months
* Chronic infectious disease, cancer, heart, kidney or liver failure;
* Pregnant, breastfeeding women or women planning a pregnancy within the year;
* Persons deprived of their liberty or subject to psychiatric care or subject to a measure of legal protection or unable to express their consent;
* Patient likely to not respect the protocol or not to be able to attend the visits, particularly given the study follow-up;
* Living at more than 30 minutes from the thermal site or who cannot be accommodated less than 30 minutes from the thermal site;
* Already included in a clinical trial or in the exclusion period of a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the eligibility criteria and living, or with possible accomodation, at less than 30 minutes from Royat (Auvergne, France)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in CIVIQ-2 score at 6 months | Baseline (D1) and final (6 months)
  The Chronic Venous Insufficiency Quality of Life Questionnaire (CIVIQ) is a disease-specific instrument to measure the impact of chronic venous insufficiency on patients' lives. CIVIQ-2 or CIVIQ-20 is a self-administered questionnaire that consists in 20 questions of the CIVIQ result in a global score. All questions have a 5-point response category, with higher scores reflecting more severe impairment. The CIVIQ-20 score ranges from 20 (minimal impact) to 100 (maximal impact).

SECONDARY OUTCOMES:
Changes from baseline in Quality of Life at 6 months | Baseline (D1) and final (6 months)
  Quality of life is measured using the generic EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state).
Changes from baseline in 0-100 VAS leg pain related to chronic venous insufficiency at 6 months | Baseline (D1) and final (6 months)
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS).
Frequency of adverse events throughout the study | From inclusion to the final visit at 6 months]
  Adverse events are described using MedDRA and each event frequency is calculated.
Participants' satisfaction with the spa therapy program at the end of the program and at 6 months | 20 days and 6 months
  Opinion of the patient is measured using a 5-point Likert scale ranging from 1 ("not at all satisfied") to 5 ("very satisfied")
Medical-economic impact of the spa therapy program at 6 months | 6 months
  EQ-5D-3L score at 6 months and frequency of adverse events related to chronic venous insufficiency.
  scores ranges from -0.541 (higher impact of health on quality of life) to 0.982 (lower impact of health on quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy COUCHET, PD, Principal Investigator — Private Practitioner
Locations (1):
- Thermes de Royat, Royat, Auvergne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier PH, Blaise S, Satger B, Genty C, Rolland C, Roques C, Bosson JL. A multicenter randomized controlled trial evaluating balneotherapy in patients with advanced chronic venous insufficiency. J Vasc Surg. 2014 Feb;59(2):447-454.e1. doi: 10.1016/j.jvs.2013.08.002. Epub 2013 Oct 15. PMID 24135621